CLINICAL TRIAL: NCT03071809
Title: Detection of Tumor DNA in Blood Samples From Patients With Early Stage Cancer and "Healthy Controls"
Status: Terminated | Type: Observational
Why Stopped: Accrual difficulties
Sponsor: Lexent Bio, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: LB-2017-03-01
Record Dates: First submitted 2017-03-01; First posted 2017-03-07 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Neoplasms, Non-hematologic - Stage I-III
Keywords: Solid tumor; carcinoma; sarcoma; stage I; stage II; stage III
MeSH Terms: conditions — Neoplasms; Carcinoma; Sarcoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood; FFPE (optional)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early stage neoplasm: Patients with stage I-III early stage non-hematologic neoplasm
- Healthy Control: Patients undergoing surgery for a non-malignant condition with no prior history of malignancy.

SUMMARY:
The aim of this study is to employ genomic detection methodologies to measure the relative amount of tumor-derived nucleic acids in the blood of patients diagnosed with an early stage solid tumor who are either commencing, currently undergoing or have completed treatment. This approach will allow the investigators to develop a quantitative measure of therapy efficacy via the counting of the relative changes in tumor molecules over the course of treatment.

DETAILED DESCRIPTION:
The aim of this study is to employ genomic detection methodologies to measure the relative amount of tumor-derived nucleic acids in the blood of patients diagnosed with an early stage solid tumor who are either commencing, currently undergoing or have completed treatment. This approach will allow the investigators to develop a quantitative measure of therapy efficacy via the counting of the relative changes in tumor molecules over the course of treatment.

The presence of circulating tumor-derived cfDNA in the plasma of patients can potentially enable a non-invasive means of detecting the presence or absence of tumor, assessing tumor burden and characterizing tumor biology in patients with cancer. The ability to measure the distribution of circulating tumor DNA may allow determination of a quantitative tumor load score in plasma that correlates to clinical tumor load. Clinical tumor load is a measure of disease burden, and the investigators propose to test in this study whether the tumor load score can measure this disease burden. A simple, reliable measure of disease burden would have diverse utility during patient therapy.

ELIGIBILITY:
Inclusion Criteria:

1. For all participants:

* Age 18 years or older
* Able to understand and grant informed consent
* Able to have their blood drawn at enrollment before surgery and 7 to 28 days after surgery

For participants with early stage solid tumors:

* Diagnosed with an early stage (I-III) solid tumor with curative intent surgery without neoadjuvant therapy planned

For "healthy control" subgroup:

* No prior or current diagnosis of any cancer. Participants with prior in situ cancer or non-melanoma skin cancer will be allowed to participate but will not be included in the "healthy control" cohort and will be analyzed separately.

Exclusion Criteria:

* Unable to grant informed consent or comply with all study procedures
* Diagnosed with a hematological malignancy (acute or chronic leukemia, myelodysplastic syndrome, myeloproliferative neoplasm, myeloma or lymphoma).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Up to 200 patients from multiple clinical sites will be enrolled in this study. Patients are eligible for this study if they are diagnosed with a solid tumor and undergoing curative resection. In addition, up to 200 participants with no prior or current diagnosis of cancer will be enrolled as a control group, i.e. "healthy control," for assay development.
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Detection of signal in the presence of active neoplasm | 2 years
  To determine the association between the tumor load score and clinical tumor load as assessed with the current standard of care methods and pathology findings.
Determine change in signal after surgery | 5 years
  To determine the response of tumor load score as a function of tumor presence as determined pre- and post-surgery intended to be curative

CONTACTS AND LOCATIONS:
Overall Officials: Haluk Tezcan, MD, Principal Investigator — Lexent Bio
Locations (1):
- Alisa Williams, MD Inc, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No